CLINICAL TRIAL: NCT02816008
Title: Smart Autonomous Neuro-Rehabilitation System
Acronym: SANaR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Pompeu Fabra (Other)
Collaborators: Hospital de la Esperanza (Unknown)
Responsible Party: Principal Investigator, Paul Verschure, PhD, Universitat Pompeu Fabra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SANaR
Record Dates: First submitted 2016-06-21; First posted 2016-06-28 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Cognition Disorders; Cognitive Deficits
Keywords: cognitive rehabilitation; memory; attention; spatial neglect; executive dysfunctioning
MeSH Terms: conditions — Cognition Disorders | interventions — PITX2 protein, human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive rehabilitation group (Experimental): Cognitive rehabilitation training with RGS in the clinic.
  Interventions: Behavioral: Cognitive rehabilitation training with RGS in the clinic
- Passive control group (Active Comparator): Passive/conventional cognitive training at home.
  Interventions: Behavioral: Passive/conventional cognitive training at home.

INTERVENTIONS:
Behavioral: Cognitive rehabilitation training with RGS in the clinic — Daily cognitive training with the Rehabilitation Gaming System (RGS) in the clinic during 6 weeks (5 days per week a 30 minutes).
  Arms: Cognitive rehabilitation group
Behavioral: Passive/conventional cognitive training at home. — Daily conventional cognitive rehabilitation at home as recommended by the neurologist during 6 weeks (5 days per week a 30 minutes).
  Arms: Passive control group

SUMMARY:
Cognitive rehabilitation is defined as a systematic functionally oriented intervention of therapeutic cognitive activities based on the assessment and understanding of patient's brain behavior deficits. This project focuses on restoring cognitive functions in order to understand the underlying deficits in the patient's brain by developing integrated cognitive rehabilitation scenarios in virtual reality that combine memory, attention and problem solving training with context specific motor movements.

ELIGIBILITY:
Inclusion Criteria:

* Score on Mini-Mental State Examination between 18 - 24
* Score on Montreal Cognitive Assessment less than 26
* More than 2 points in upper limb motor scale MRC
* Sufficient cognitive ability to understand and follow the experimental instructions

Exclusion Criteria:

* Score on Mini-Mental State Examination below 18 or above 24
* Score on Montreal Cognitive Assessment of 26 or above
* Below 2 point in upper limb motor scale MRC
* Hemianopia
* Cognitive capacity that prohibits the execution of the experiment
* Severe impairment like spasticity, aphasia or apraxia, major pain or other neuromuscular impairments or dependent on use of orthopedic devices that would interfere with the correct execution of understanding of the experiment
* History of serious mental-health problems in acute or subacute phase
* Patients that do not give their consent to participate in the study

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-07; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change in Digit Span Forward WAIS-IV from baseline to end of treatment and to follow-up | Measured at baseline, at 6 weeks (end of treatment), and at 3-months (follow-up)
  Measurement of attention
Change in Corsi block tapping test from baseline to end of treatment and to follow-up | Measured at baseline, at 6 weeks (end of treatment), and at 3-months (follow-up)
  Measurement of attention
Change in Trail Making Test, Part A from baseline to end of treatment and to follow-up | Measured at baseline, at 6 weeks (end of treatment), and at 3-months (follow-up)
  Measurement of attention
Change in Rey Auditory Verbal Learning Test from baseline to end of treatment and to follow-up | Measured at baseline, at 6 weeks (end of treatment), and at 3-months (follow-up)
  Measurement of episodic memory
Change in Digit Span Backward WAIS-IV from baseline to end of treatment and to follow-up | Measured at baseline, at 6 weeks (end of treatment), and at 3-months (follow-up)
  Measurement of working memory
Change in Corsi block-tapping test reversed from baseline to end of treatment and to follow-up | Measured at baseline, at 6 weeks (end of treatment), and at 3-months (follow-up)
  Measurement of working memory
Change in Frontal Assessment Battery from baseline to end of treatment and to follow-up | Measured at baseline, at 6 weeks (end of treatment), and at 3-months (follow-up)
  Measurement of executive functioning
Change in Trail Making Test, Part B from baseline to end of treatment and to follow-up | Measured at baseline, at 6 weeks (end of treatment), and at 3-months (follow-up)
  Measurement of set-shifting
Change in Digit Symbol Coding in WAIS-IV from baseline to end of treatment and to follow-up | Measured at baseline, at 6 weeks (end of treatment), and at 3-months (follow-up)
  Measurement of processing speed
Change in Star Cancellation test from baseline to end of treatment and to follow-up | Measured at baseline, at 6 weeks (end of treatment), and at 3-months (follow-up)
  Measurement of spatial neglect

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment from baseline to end of treatment and to follow-up | Measured at baseline, at 6 weeks (end of treatment), and at 3-months (follow-up)
  Measurement of global cognitive ability
Change in Mini-Mental State Examination from baseline to end of treatment and to follow-up | Measured at baseline, at 6 weeks (end of treatment), and at 3-months (follow-up)
  Measurement of global health status
Change in Barthel Index from baseline to end of treatment and to follow-up | Measured at baseline, at 6 weeks (end of treatment), and at 3-months (follow-up)
  Measurement of independent functioning and mobility in activities of daily living
Change in Fugl-Meyer Assessment from baseline to end of treatment and to follow-up | Measured at baseline, at 6 weeks (end of treatment), and at 3-months (follow-up)
  Measurement of motor recovery after stroke

CONTACTS AND LOCATIONS:
Overall Officials: Esther Duarte Oller, MD, PhD, Principal Investigator — Parc de Salut Mar - Hospital de l'esperança; Paul F.M.J. Verschure, PhD, Study Director — Director Specs

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cicerone KD, Langenbahn DM, Braden C, Malec JF, Kalmar K, Fraas M, Felicetti T, Laatsch L, Harley JP, Bergquist T, Azulay J, Cantor J, Ashman T. Evidence-based cognitive rehabilitation: updated review of the literature from 2003 through 2008. Arch Phys Med Rehabil. 2011 Apr;92(4):519-30. doi: 10.1016/j.apmr.2010.11.015. PMID 21440699
- [Background] Ball K, Berch DB, Helmers KF, Jobe JB, Leveck MD, Marsiske M, Morris JN, Rebok GW, Smith DM, Tennstedt SL, Unverzagt FW, Willis SL; Advanced Cognitive Training for Independent and Vital Elderly Study Group. Effects of cognitive training interventions with older adults: a randomized controlled trial. JAMA. 2002 Nov 13;288(18):2271-81. doi: 10.1001/jama.288.18.2271. PMID 12425704
- [Background] Corbetta M, Ramsey L, Callejas A, Baldassarre A, Hacker CD, Siegel JS, Astafiev SV, Rengachary J, Zinn K, Lang CE, Connor LT, Fucetola R, Strube M, Carter AR, Shulman GL. Common behavioral clusters and subcortical anatomy in stroke. Neuron. 2015 Mar 4;85(5):927-41. doi: 10.1016/j.neuron.2015.02.027. PMID 25741721
- [Background] Nair RD, Lincoln NB. Cognitive rehabilitation for memory deficits following stroke. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD002293. doi: 10.1002/14651858.CD002293.pub2. PMID 17636703
- [Derived] Maier M, Ballester BR, Leiva Banuelos N, Duarte Oller E, Verschure PFMJ. Adaptive conjunctive cognitive training (ACCT) in virtual reality for chronic stroke patients: a randomized controlled pilot trial. J Neuroeng Rehabil. 2020 Mar 6;17(1):42. doi: 10.1186/s12984-020-0652-3. PMID 32143674